CLINICAL TRIAL: NCT01819974
Title: Effect of Medication Reviews in Hospitalized High-risk Patients - a Randomised Controlled Trial
Brief Title: Effect of Medication Reviews Performed in High Risk Patients
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: University of Aarhus (Other)
Collaborators: Aarhus University Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: MERIS2
Record Dates: First submitted 2013-03-18; First posted 2013-03-28 (Estimated); Last update posted 2013-11-28 (Estimated); Status verified 2013-11

CONDITIONS: Patients in Highest Medication Error Risk

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Control (No Intervention): The normal procedure at the ward
- Stratified medication review (Active Comparator): Medication review performed by either a clinical pharmacist or a clinical pharmacologist in patients with highest medication error risk
  Interventions: Other: Stratified medication review

INTERVENTIONS:
Other: Stratified medication review — A mediciation review will be performed in patients with high medication error rik. Patients in the highest risk will receive the medication review from a clinical pharmacologist whereas patients assessed in lesser risk will receive the medication review from a clinical pharmacist.
  Arms: Stratified medication review

SUMMARY:
The purpose of the study is to examine whether a stratified medication review performed in patients at highest risk of experiencing medication errors have impact on numbers of medication errrors during hospitalization.

DETAILED DESCRIPTION:
Acutely admitted medical patients will be included after admission. After inclusion and randomization the patients will be risk stratified with an existing algorithm according to risk of medication error. The patients in the intervention group will receive a medication review performed by a clinical pharmacist if they are in high medication error risk. Patients in highest medication error risk will recieve a medication review performed by a clinical pharmacologist.

ELIGIBILITY:
Inclusion Criteria:

* Acutely admitted
* >17 years
* Patients being treated with at least one drug at admission

Exclusion Criteria:

* Dying patients
* Suicidal patients
* Intoxicated patients

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 600 (Estimated)
Dates: Start 2013-04; Primary Completion 2013-11 (Estimated); Study Completion 2014-05 (Estimated)

PRIMARY OUTCOMES:
Medication errors | During hospitalization ie. between 8 hours and approximately 20 days
  Medication errors are defined as errors in prescribing that has the potential to harm patients or actually harm patients. This will be assessed by checking the medical records. Two independent experts will do this.

SECONDARY OUTCOMES:
hospital readmissions (all-cause) | 3 months after discharge

CONTACTS AND LOCATIONS:
Locations (1):
- Aarhus University Hospital, Aarhus, Denmark